CLINICAL TRIAL: NCT02768610
Title: Effects of Preanesthetic Dexmedetomidine on Hemodynamic Responses to Endotracheal Intubation in Elderly Patients Being Treated for Hypertension: A Randomized Trial
Brief Title: Use of Preanesthetic Dexmedetomidine in Elderly, Treated-hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Chanwoo Lee, M.D., DongGuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 110757-201602-HR-03-03
Record Dates: First submitted 2016-05-05; First posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Perioperative Care
Keywords: dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- dexmedetomidine (Experimental): 0.5 mcg/kg dexmedetomidine is administered before endotracheal intubation for 10 minutes
  Interventions: Drug: Dexmedetomidine
- Normal Saline (Placebo Comparator)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: dexmedetomidine
Drug: Normal Saline
  Arms: Normal Saline

SUMMARY:
Background: Dexmedetomidine is an alpha 2 adrenergic agonist with sedative, anxiolytic, and analgesic properties. This study was designed to evaluate the inhibitory effects of preoperative 0.5 μg/kg dexmedetomidine on hemodynamic responses caused by endotracheal intubation in elderly patients being treated for hypertension.

Methods: Forty elderly (≥ 65 years) treated-hypertensive patients of American Society of Anesthesiologists physical status II undergoing elective noncardiac surgery were randomly and assigned to two groups. Group C received normal saline and group D received 0.5 μg/kg dexmedetomidine intravenously over 10 min just before endotracheal intubation. Systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP) and heart rate (HR) were recorded preoperatively at ward, immediately after study drug administration, and at 1, 3, and 5 minutes after endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status II
* Scheduled for elective noncardiac surgery
* Being treated with anti-hypertensive medication

Exclusion Criteria:

* Endotracheal intubation attempted more than twice
* Morbidly obese (BMI > 35 kg/m2)

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes in systolic blood pressure | 2 minutes before intubation and 1, 3, 5 minutes after intubation
  Units of Measure : mmHg
Changes in diastolic blood pressure | 2 minutes before intubation and 1, 3, 5 minutes after intubation
  Units of Measure : mmHg
Changes in mean arterial pressure | 2 minutes before intubation and 1, 3, 5 minutes after intubation
  Units of Measure : mmHg
Changes in heart rate | 2 minutes before intubation and 1, 3, 5 minutes after intubation
  Units of Measure : beats/min

CONTACTS AND LOCATIONS:
Overall Officials: Miwoon Kim, M.D., Ph.D., Study Director — DongGuk universit hospital Gyeongju hospital